CLINICAL TRIAL: NCT02434224
Title: Creative Music Therapy for Premature Infants: Testing a Possible Influence on Brain Structure, Function and Neurobehavioral Outcome
Brief Title: Creative Music Therapy for Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-0655
Record Dates: First submitted 2015-03-30; First posted 2015-05-05 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Developmental Delay (Disorder)
Keywords: Music therapy; premature infant; brain development
MeSH Terms: conditions — Developmental Disabilities; Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- music therapy (Experimental): two to three sessions per week: The therapist will stay with one hand on the infants' chest (or back) in order to continuously assess the infants' breathing pattern. Based on and oriented towards the assessed breathing pattern, the infants' behavioral state, facial and gestural expression, the therapist transforms the infants' rhythms and subtle expressions into infant-directed improvised humming.
  Interventions: Procedure: Music Therapy
- control (No Intervention): standard care

INTERVENTIONS:
Procedure: Music Therapy — 2 to 3 sessions per week of individualized creative music therapy
  Arms: music therapy

SUMMARY:
This study investigates whether creative music therapy applied to premature infants will facilitate brain growth and development at term equivalent assessed by magnetic resonance imaging. Secondary objective are improvement of neurobehavioral outcomes of premature infants at 24 months, as well as at 5 years of age.

DETAILED DESCRIPTION:
Premature infants are a highly prevalent and vulnerable group in paediatric care, and face several short- and long-term challenges. Research on brain development in premature infants demonstrates a high incidence of white and grey matter abnormalities and neurobehavioral delay, as well as an increased risk of brain injury. There is growing awareness that premature infants need individualized nurturing interactions with their caregivers while they are in a neonatal intensive care unit (NICU) to support healthy development and prevent future difficulties. One particular intervention that may have considerable potential in the NICU is creative music therapy (CMT), an individualized, interactive, resource- and needs-oriented music therapy approach. Results demonstrate that CMT can facilitate relaxation and stabilization in premature infants; by experiencing inter-subjectivity through music, the infants can be empowered to engage in meaningful and nurturing interactions (Haslbeck, 2013 a,b) .

Several researchers (Als, 2012; Trevarthen, 2008; Schore, 2003) have described how interactive and multi-sensory experiences of the fetus particularly facilitate brain development and learning about socio-emotional figures, respectively, in prematurely born infants. It is assumed that positive auditory experiences can promote premature infants' early brain maturation and contribute to their healthy neurodevelopment (Xu et al., 2009). Studies in music and neuroscience have demonstrated that music promotes neurobiological processes and modulates synaptic plasticity, neuronal learning and readjustment in the human brain (Rickard et al., 2005). The individualized approach in active music therapy may especially activate brain structures involved in emotional, sensorimotor and cognitive processing (Koelsch, 2009; Fachner et al., 2012).

Since, on one hand, individualized interactive experiences and, on the other hand, music may alter brain development in the fetus and very young infants, the question arises as to whether CMT might actually promote a premature infant's brain development by facilitating nurturing socio-emotional and auditory interactive experiences at the same time. Therefore a randomized, controlled, clinical trial will be conducted. 30 premature infants receive CMT during their hospitalization time and 30 premature infants without music therapy serves as control group. The primary objective is to explore if the experience of CMT in premature infants improves their brain growth and development at 38-42 weeks of corrected gestational age. The main secondary objective is to explore if CMT improves the neurobehavioral outcomes of premature infants at 9 and 24 months, as well as at 5 years of age. Magnetic resonance imaging is used to evaluate the infants' cerebral cortical development and myelination. Electroencephalography (EEG) is used to evaluate the infants' brain function and maturation. Insights into possible long-term and sustainable outcomes will be gained via neuro-developmental follow-up examinations. It is hypothesized that the experience of CMT in neonatal care improves both short- and long-term neurological outcomes. We expect that the experimental group will demonstrate superior brain growth and development at 38-42 weeks of corrected gestational age as well as improved cognitive, behavioral and motor developmental outcomes later on. This paper will introduce first insights and preliminary results of the ongoing study. Strategies and challenges inherent in conducting a controlled clinical trial within this vulnerable group will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Born before 32 weeks of gestational age
* Clinically stable
* Chronological age ≥ 7 days of life
* Informed written parental consent

Exclusion Criteria:

* Born after 32 weeks of gestational age (due to a possible too short timeframe for music therapy treatment)
* Lack of parental consent
* Admitted a priori for palliative care
* Genetically defined syndrome
* Severe congenital malformation adversely affecting life expectancy or neurodevelopment
* (For the control group only: Regular singing or other kinds of music stimulation by the parents during hospitalization time)

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Brain volume | 40 gestational weeks
  3D magnetic resonance volumetric analysis: volumes of white matter (myelinated and unmyelinated) and grey matter volume will be evaluated

SECONDARY OUTCOMES:
Mental Development Index (Bayley III) | 24 months corrected for prematurity
  Bayley scales III (MDI)
Intelligence Quotient | 5 years
  Intelligence quotient (Wechsler Preschool and Primary Scale of Intelligence-Revised, WPPSI-R) to determine long-term development and intelligence. Children will be classified as either being normal or having minor or major impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Hans U Bucher, Prof., Study Chair — University of Zurich
Locations (1):
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Haslbeck FB, Bucher HU, Bassler D, Hagmann C, Natalucci G. Creative Music Therapy and Neurodevelopmental Outcomes in Pre-term Infants at 2 Years: A Randomized Controlled Pilot Trial. Front Pediatr. 2021 Jun 18;9:660393. doi: 10.3389/fped.2021.660393. eCollection 2021. PMID 34222141
- [Derived] Haslbeck FB, Bucher HU, Bassler D, Hagmann C. Creative music therapy to promote brain structure, function, and neurobehavioral outcomes in preterm infants: a randomized controlled pilot trial protocol. Pilot Feasibility Stud. 2017 Sep 26;3:36. doi: 10.1186/s40814-017-0180-5. eCollection 2017. PMID 28975039